CLINICAL TRIAL: NCT02721199
Title: Investigation of Factors Affecting Respiratory Muscle EMG Measurements During Hospital Admission With Acute Exacerbation of COPD
Brief Title: EMG in COPD - Factor Analysis
Acronym: EMGCOPD
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 178765
Record Dates: First submitted 2016-01-27; First posted 2016-03-29 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prospective Cohort: Neural Respiratory Drive Automated EMGpara assessment
  Interventions: Other: Neural Respiratory Drive Automated EMGpara assessment

INTERVENTIONS:
Other: Neural Respiratory Drive Automated EMGpara assessment — Neural respiratory drive will be measured using surface electrodes and nasal cannula . The 2nd intercostal space will be identified by bony landmarks and skin preparation will be performed using detergent wipes, followed by EMG preparation gel with final cleaning to remove exfoliated skin. Wet gel electrodes will be placed immediately adjacent to the sternal border in the 2nd intercostal space and will be connected to the automated EMG analysis system. Electrodes will remain in place for the duration of the study. A nasal cannula will be placed in the nose and detect pressure changes during respiration in order to ensure accurate detection of inspiratory cycle. In addition, an accelerometer will be attached to the thorax of the patient

SUMMARY:
Acute exacerbations of COPD contribute to significant morbidity and mortality in the United Kingdom (UK). The ability to assess response to treatment during exacerbations that require hospitalisation would allow clinicians to better risk stratify patients for higher or lower level in-patient or out-patient care. Current methods of detecting clinical deterioration are validated in general medical populations and may lack sensitivity and specificity in patients with respiratory morbidity. The use of respiratory muscle EMG to assess neural respiratory drive (NRD) has been demonstrated to be a predictor of readmission in patients admitted to hospital with COPD. The technique has been applied on 'spot' readings of limited duration due to the need for hand analysis of the data. It has been performed by a trained clinical physiologist who removed any interference data and standardised the data gathered. New automated software allows for longer periods of observation, mostly unsupervised, and as a result, the NRD measurements are more likely to be affected by various sources of variability. The influence of clinical and physiological factors as they occur during routine clinical management, such as administration of bronchodilator medication, time of day of readings or proximity to chest physiotherapy, are not yet understood. This trial is designed to gather data to better understand these relationships with NRD.

DETAILED DESCRIPTION:
Introduction Patients admitted to hospital with acute exacerbations of COPD are at risk of significant in-hospital morbidity and mortality. Current markers of treatment success involve the integration of basic physiological variables (respiratory rate, heart rate, oxygen saturations), clinical examination and patient reported symptoms changes. Whilst the use of these physiological parameters are gold standard there remains concern that patient deterioration is often not detected and escalated effectively. This has led to the development and implementation of a range of clinical physiological composite scores such as the medical early warning score or the National Health Service (NHS) early warning scores. However, these scores have been validated in general rather than specific populations and there are concerns regarding their use in respiratory patient groups.The use of the parasternal intercostal muscle EMG (EMGpara) has been reported to track clinical change and identify treatment failure during hospital admissions with acute exacerbations of COPD (AECOPD) in selected and unselected cohorts. In these pilot works measurements were taken on research equipment and data analysed individually by a trained physiologist. The clinical physiologist ensured standardisation of recording conditions such as proximity to medication, patient position, time of day and recent activity. The effect of such clinical and physiological factors on EMGpara was minimised by the operator with preventive measures, such as the control for the measurement time, the limitation of the recording duration and the exclusion of any artefactual changes in EMGpara. The development of automated software allows for frequent sampling and continuous monitoring, which will potentially permit earlier detection of clinical deterioration. With an automated system however, clinical and physiological factors need to be carefully considered, in particular when the measurement is performed in an unsupervised or less closely supervised environment. This feasibility study is therefore designed to investigate repeatability of EMGpara in hospital-based AECOPD management (i.e. EMGpara changes reflect changes in clinical status). It will give us insight into potential control/mitigation measures and their implementation, in order to ultimately minimise false readings.

Study objectives To investigate the clinical and physiological factors that may affect the measurement of EMGpara in acute setting so as to enhance the clinical effectiveness of EMGpara in identifying treatment failure and clinical deterioration.

ELIGIBILITY:
Inclusion Criteria:

* COPD (as defined by GOLD criteria
* Acute exacerbation of COPD necessitating hospital admission
* Expected to remain an inpatient for ≥ 24 hours
* Able to give informed consent to participation in the study

Exclusion Criteria:

* Decompensated respiratory failure (pH < 7.35)
* Significant physical, social or psychiatric factors that would prevent compliance with trial protocol
* Aged < 35 years or aged > 85 years
* Pregnancy
* BMI > 30kg/m2
* Presence of another acute pathology (such as pulmonary embolism or pulmonary oedema) to explain the acute presentation

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to St Thomas' Hospital with a primary diagnosis of an acute exacerbation of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting Medication Intake | 3 days
  Noting all medications taken during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting oxygen therapy. | 3 days
  Noting oxygen therapy, if any during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting use of non invasive ventilation. | 3 days
  Noting use of non invasive ventilation, if any during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting intubation details. | 3 days
  Noting details if participant is intubated during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting information if participant is transferred to critical care. | 3 days
  Noting details if participant is transferred to critical care during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting information if participant takes part in a respiratory physiotherapy session. | 3 days
  Noting details if participant takes part in a respiratory physiotherapy session during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), physiological factors that change EMG parasternal readings. If participant goes into clinical respiratory deterioration by the need for treatment/care escalation. | 3 days
  Noting details if participant is intubated during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of COPD, the physiological factors that can change EMG parasternal readings. If participant goes into clinical respiratory deterioration National Early Warning Score (NEWS) CREWS | 3 days
  Noting details if participant is documented as being in clinical respiratory deterioration as defined by NEWS/CREWS during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting information if participant partakes in physical activity | 3 days
  Noting details if participant partakes in any physical activity during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), physiological factors that change EMG parasternal readings. Collecting information when participant sleeps | 3 days
  Noting details when participant sleeps during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting information if there is any postural change | 3 days
  Noting details if participant changes postural position during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day.
During the course of an exacerbation of Chronic Obstructive Pulmonary Disease (COPD), the physiological factors that can change EMG parasternal readings. Collecting information if participant takes part in a rehabilitation physiotherapy session. | 3 days
  Noting details if participant takes part in a rehabilitation physiotherapy session during the time frame up to 3 days during the exacerbation of COPD. Information taken 4 times during the day at the same time each day

SECONDARY OUTCOMES:
Is it possible to perform Continuous EMGpara acquisition in a clinical setting | 3 Days
Continuous EMGpara acquisition in clinical setting, is it applicable. | 3 Days
Continuous EMGpara acquisition in clinical setting, preliminary insights on device requirements for this environment. | 3 Days
EMGpara trends as it relates to standardly used metrics, e.g. vital signs, patient-reported symptoms. | 3 Days
Rhe automated neural respiratory drive (NRD) calculation algorithm during continuous measurements will be optimised to increase the robustness of the algorithm against artefacts. | 3 Days
Standardise the measurement set-up and measurement protocol in routine AECOPD management. | 3 Days

CONTACTS AND LOCATIONS:
Overall Officials: Nick Hart, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No